CLINICAL TRIAL: NCT05985265
Title: Assessment of Nano Fat Grafting Combined With Fractional Carbon Dioxide Laser Resurfacing Versus Nano Fat Grafting Alone in Atrophic Facial Acne Scars
Brief Title: Nano Fat Injection With or Without Fractional Carbon Dioxide Laser in Acne Scars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Hisham Zayan, resident plastic surgery department, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: nano fat injection
Record Dates: First submitted 2022-11-15; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Acne Scars - Atrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nano fat grafting and fractional carbon dioxide laser resurfacing (Experimental): treating of atrophic acne scars with nano fat and fractional carbon dioxide laser
  Interventions: Procedure: Fat grafting

INTERVENTIONS:
Procedure: Fat grafting — Nano fat grafting followed by fractional carbon dioxide laser resurfacing
  Other Names: fractional carbon dioxide laser resurfacing

SUMMARY:
Assessment of nano fat grafting combined with carbon dioxide laser resurfacing versus nano fat grafting alone in treating facial atrophic acne scars

DETAILED DESCRIPTION:
Acne scars is a world wide problem .though lots of treatment exists still mo gold standard for treatment of acne scars in this study.

Assessment of nano fat grafting combined with carbon dioxide laser resurfacing versus nano fat grafting alone in treating facial atrophic acne scars

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years who attend the Outpatient Clinics of Dermatology and Plastic Surgery Departments, Assiut University Hospital, with moderate to severe atrophic facial acne scars on both cheeks, as assessed using the Goodman and Baron Qualitative scar grading system (12), will be enrolled in the study.

Exclusion Criteria:

* include: pregnancy or lactation; active acne, history of deep chemical peeling or filler injection in the previous 6 months, history of keloid or hypertrophic scar formation; use of isotretinoin in the previous 6 months; active infection in the treatment area; bleeding tendencies; history of herpes simplex or herpes zoster infection on the face; and patients with unrealistic expectations.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-04-29 (Estimated); Study Completion 2024-05-29 (Estimated)

PRIMARY OUTCOMES:
Clinical assessment of acne scar severity | up to 24 weeks
  as assessed using the Goodman and Baron Qualitative scar grading system before and after treatment on both sides of face, to determine the number of patients achieving two grades improvement vs one grade or no improvement

SECONDARY OUTCOMES:
Physician global assessment | up to 24 weeks
  two blinded observers will compare the before and after photographs separately on each facial side and will evaluate the improvement on a quartile grading scale as: poor,<25% improvement; fair, 25%-50% improvement; good, 51%-75% improvement; and excellent, >75% improvement.
percent of reduction in scar count | up to 24 weeks
  count of the total and different types of acne scars was performed, before and after treatment on both sides of the face, and the percent of reduction was calculated
Patient satisfaction | 1 year
  Patients will rate their overall satisfaction on a quartile grading system: 0, unsatisfied; 1, slightly satisfied; 2, satisfied; and 3, very satisfied
Adverse events | 1 year
  erythema, edema, crusting, pigmentary changes, ecchymosis, and scarring, will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: youssef S farrag, MD, Principal Investigator — Department of Plastic Surgery, professor; Wael S Ibraheem, MD, Principal Investigator — Department of Plastic Surgery , Assistant lecture
Locations (1):
- Faculty of Medicine, Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goodman GJ, Baron JA. Postacne scarring: a qualitative global scarring grading system. Dermatol Surg. 2006 Dec;32(12):1458-66. doi: 10.1111/j.1524-4725.2006.32354.x. PMID 17199653
- [Result] Jacob CI, Dover JS, Kaminer MS. Acne scarring: a classification system and review of treatment options. J Am Acad Dermatol. 2001 Jul;45(1):109-17. doi: 10.1067/mjd.2001.113451. PMID 11423843
- [Result] Chan NP, Ho SG, Yeung CK, Shek SY, Chan HH. Fractional ablative carbon dioxide laser resurfacing for skin rejuvenation and acne scars in Asians. Lasers Surg Med. 2010 Nov;42(9):615-23. doi: 10.1002/lsm.20974. PMID 20976801